CLINICAL TRIAL: NCT04738994
Title: Effects of Whey Protein-enriched Nutritional Supplement on Gut Microbiota and Inflammatory Status, in Patients Attending a Cardiac Rehabilitation Program
Brief Title: Nutritional Support for Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other); University of Florence (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: wheyprotein1_FDG
Record Dates: First submitted 2021-02-02; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Rehabilitation
Keywords: whey protein; gut microbiota; interleukin 6; cardiac rehabilitation; nutritional supplement; inflammatory status
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whey protein-enriched nutritional supplement (Experimental): Standard hospital diet + 80 g/die (two servings) of whey protein-enriched nutritional supplement dissolved in 125 ml of water
  Interventions: Dietary Supplement: whey protein-enriched nutritional supplement
- Control group (Active Comparator): Standard hospital diet
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: whey protein-enriched nutritional supplement — Standard hospital diet + 80 g/die (two servings) of whey protein-enriched nutritional supplement dissolved in 125 ml of water
  Arms: whey protein-enriched nutritional supplement
Other: Control group — Standard hospital diet
  Arms: Control group

SUMMARY:
In this randomized trial the primary outcome is to assess if high doses of whey protein supplement may lower pro-inflammatory interleukin 6 (IL-6).

Hypothesis: Secondary outcomes are to assess if high doses of whey protein supplement may lower pro-inflammatory interleukin 1β (IL-1 β), tumor necrosis factor and C Reactive Protein (CRP); may increase anti-inflammatory interleukin 10 (IL-10) plasma concentrations and may change Gut Microbiota (GM) composition.

ELIGIBILITY:
Inclusion Criteria:

* Admission for cardiac rehabilitation
* Signed informed consent

Exclusion Criteria:

* Patient unable to eat orally
* Eating disorders
* Indication to Levodopa therapy
* Gastrointestinal malignant diseases
* Known kidney failure
* Known liver failure
* Previous antibiotic therapy
* Refusal

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pro-inflammatory cytokine interleukin 6 (IL-6) | Baseline (T0) and day 15 (T1)
  Change in IL-6 [Time Frame: after 15 days (T1) from baseline (T0)]

SECONDARY OUTCOMES:
Pro-inflammatory cytokine interleukin 1beta (IL-1β) | Baseline (T0) and day 15 (T1)
  Change in IL-1β [Time Frame: after 15 days (T1) from baseline (T0)]
Tumor Necrosis Factor (TNF) | Baseline (T0) and day 15 (T1)
  Change in TNF [Time Frame: after 15 days (T1) from baseline (T0)]
C-Reactive Protein (CRP) | Baseline (T0) and day 15 (T1)
  Change in CRP [Time Frame: after 15 days (T1) from baseline (T0)]
Anti- inflammatory cytokine interleukin 10 (IL-10) | Baseline (T0) and day 15 (T1)
  Change in IL-10 [Time Frame: after 15 days (T1) from baseline (T0)]
Gut Microbiota (GM) | Baseline (T0) and day 15 (T1)
  Change in GM [Time Frame: after 15 days (T1) from baseline (T0)]

CONTACTS AND LOCATIONS:
Overall Officials: Chiara F Gheri, MD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus
Locations (1):
- Fondazione Don Carlo Gnocchi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Aguilar-Nascimento JE, Prado Silveira BR, Dock-Nascimento DB. Early enteral nutrition with whey protein or casein in elderly patients with acute ischemic stroke: a double-blind randomized trial. Nutrition. 2011 Apr;27(4):440-4. doi: 10.1016/j.nut.2010.02.013. Epub 2010 Dec 16. PMID 21167685
- [Background] Sugawara K, Takahashi H, Kashiwagura T, Yamada K, Yanagida S, Homma M, Dairiki K, Sasaki H, Kawagoshi A, Satake M, Shioya T. Effect of anti-inflammatory supplementation with whey peptide and exercise therapy in patients with COPD. Respir Med. 2012 Nov;106(11):1526-34. doi: 10.1016/j.rmed.2012.07.001. Epub 2012 Aug 3. PMID 22857881
- [Background] Zhou LM, Xu JY, Rao CP, Han S, Wan Z, Qin LQ. Effect of whey supplementation on circulating C-reactive protein: a meta-analysis of randomized controlled trials. Nutrients. 2015 Feb 9;7(2):1131-43. doi: 10.3390/nu7021131. PMID 25671415
- [Background] Fekete AA, Givens DI, Lovegrove JA. Can milk proteins be a useful tool in the management of cardiometabolic health? An updated review of human intervention trials. Proc Nutr Soc. 2016 Aug;75(3):328-41. doi: 10.1017/S0029665116000264. Epub 2016 May 6. PMID 27150497
- [Background] Laviolette L, Lands LC, Dauletbaev N, Saey D, Milot J, Provencher S, LeBlanc P, Maltais F. Combined effect of dietary supplementation with pressurized whey and exercise training in chronic obstructive pulmonary disease: a randomized, controlled, double-blind pilot study. J Med Food. 2010 Jun;13(3):589-98. doi: 10.1089/jmf.2009.0142. PMID 20521985
- [Background] Kerasioti E, Stagos D, Jamurtas A, Kiskini A, Koutedakis Y, Goutzourelas N, Pournaras S, Tsatsakis AM, Kouretas D. Anti-inflammatory effects of a special carbohydrate-whey protein cake after exhaustive cycling in humans. Food Chem Toxicol. 2013 Nov;61:42-6. doi: 10.1016/j.fct.2013.01.023. Epub 2013 Jan 27. PMID 23360676